CLINICAL TRIAL: NCT03007966
Title: Ilioinguinal/Iliohypogastric vs. Quadratus Lumborum Nerve Blockade for Elective Open Inguinal Herniorrhaphy
Brief Title: IINB vs. QLB for Elective Open Inguinal Herniorrhaphy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00040354
Record Dates: First submitted 2016-12-22; First posted 2017-01-02 (Estimated); Results first posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-10

CONDITIONS: Nerve Block; Herniorrhaphy; Regional Anesthesia
MeSH Terms: interventions — Epinephrine; Clonidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ilioinguinal / Iliohypogastric Block (Active Comparator): Patient's randomized to receive an Ilioinguinal / Iliohypogastric nerve block (IINB) for post operative analgesia following inguinal herniorrhaphy will have said block performed in a supine position in a manner consistent with the technique described by Willschke, but modified to utilize an in-plane technique rather than an out-of-plane technique for needle to ultrasound probe orientation. Either a Sonosite linear HFL38x/13-6 MHz or Sonosite curvilinear C60x/5-2 MHz probe will be utilized to visualize the pertinent ultrasound anatomy. A Pajunk 21g x 100mm Sono Plex Stim Cannula will be utilized to appropriately deposit a single local anesthetic aliquot consisting of 25cc's of bupivacaine 0.25% with epinephrine 5mcg/cc and clonidine 1.66mcg/cc.
  Interventions: Procedure: Ilioinguinal / Iliohypogastric Block; Drug: Bupivacaine 0.25%; Drug: Epinephrine 1:200k; Drug: Clonidine 1.66mcg/cc
- Quadratus Lumborum Block (Experimental): Patient's randomized to receive a Quadratus Lumborum block (QLB) for post operative analgesia following inguinal herniorrhaphy will have said block performed in a lateral position in a manner consistent with the technique described by Børglum. Either a Sonosite linear HFL38x/13-6 MHz or Sonosite curvilinear C60x/5-2 MHz probe will be utilized to visualize the pertinent ultrasound anatomy. A Pajunk 21g x 100mm Sono Plex Stim Cannula will be utilized to appropriately deposit a single local anesthetic aliquot consisting of 25cc's of bupivacaine 0.25% with epinephrine 5mcg/cc and clonidine 1.66mcg/cc.
  Interventions: Procedure: Quadratus Lumborum Block; Drug: Bupivacaine 0.25%; Drug: Epinephrine 1:200k; Drug: Clonidine 1.66mcg/cc

INTERVENTIONS:
Procedure: Ilioinguinal / Iliohypogastric Block — Patients randomized to this arm will receive 25cc's of Bupivacaine 0.25% + Epinephrine 1:200k + Clonidine 1.66mcg/cc administered via an ultrasound guided ilioinguinal / iliohypogastric block technique.
  Arms: Ilioinguinal / Iliohypogastric Block
Procedure: Quadratus Lumborum Block — Patients randomized to this arm will receive 25cc's of Bupivacaine 0.25% + Epinephrine 1:200k + Clonidine 1.66mcg/cc administered via an ultrasound guided quadratus lumborum block technique.
  Arms: Quadratus Lumborum Block
Drug: Bupivacaine 0.25% — Administered as part of the local anesthetic mixture
Drug: Epinephrine 1:200k — Administered as part of the local anesthetic mixture
Drug: Clonidine 1.66mcg/cc — Administered as part of the local anesthetic mixture

SUMMARY:
Open inguinal herniorrhaphy is a common outpatient surgical procedure. Post-operative pain can be a significant hindrance to discharge from the post anesthesia care unit. Pain can be treated with opioid therapy, but the literature supports that these agents are known to create or exacerbate adverse effects and complications, including post-operative nausea and vomiting, hypoxia, and urinary retention. In contrast, analgesia provided by regional anesthesia results in a decreased risk of the aforementioned complications.1 Because of this, various regional anesthetic techniques have been developed to provide analgesia following open herniorrhaphy. One technique is a combined ilioinguinal and iliohypogastric nerve block (IINB), which has been shown to decrease the initial pain after inguinal herniorrhaphy.2 The quadratus lumborum block (QLB) is a newer regional anesthetic technique that we think could be as effective as IINB at providing pain control following open herniorrhaphy. Additionally, because local anesthetic injected during a QLB has the potential to spread cranially into the thoracic paravertebral space following its lumbar deposition it could lead to alleviation of both somatic and visceral pain.3 This might therefore improve the quality and or duration of analgesia as compared to the IINB. To the best of the author's knowledge there has been no investigation comparing the efficacy, with regards to post-operative pain management, between IINB and QLB.

DETAILED DESCRIPTION:
This study will be a double-blinded prospective randomized controlled equivalency trial comparing QLB to IINB. Patients presenting for unilateral open inguinal herniorrhaphy who agree to participate in the study and do not meet exclusion criteria will be randomized to either receiving an IINB or a QLB for post-operative analgesia. After performing a timeout, applying monitors (ECG, capnography, Sp02, non-invasive blood pressure), and confirming all paperwork per the usual pre-procedural check list the study participants will be administered procedural sedation (fentanyl and midazolam) to comfort as well as supplemental oxygen. The anatomy of both block sites will be identified by palpation of landmarks, labeling of structures with a skin marking pen, and visualization under ultrasound guidance. Both sites will be administered a small skin wheal of lidocaine 1% at the site the block needle would be introduced into the skin. Our intent with regards to administering a local anesthetic skin wheal is to increase our success in blinding the patient to which block was actually performed. A regional anesthetic block will only be performed at the randomized block site (IINB vs. QLB). After 15-30 minutes post block or post operatively the block will be assessed for success. Loss of cold sensation in the area of the surgical site would be indicative of block success. The patient will then proceed to the operating room and receive a general anesthetic with the final details of that anesthetic to be determined by the anesthesiologist responsible for the patient in the operating room. We will ask the operating room anesthesiologist and surgeon to avoid administration of medications that would confound our results. Specifically, no additional local anesthetic is to be injected at the incision site, no long acting opioids (hydromorphone, morphine, methadone etc…), dexamethasone or ketamine. After completion of the procedure the patient will recover in the post anesthesia care unit (PACU) where the participant will recover as per the usual process. The patient's discharge disposition will be at the discretion of the surgeon and anesthesiologist responsible for the participant's PACU care. The patient will be provided a diary that the participant will complete at 8hrs and 24hrs post block that will help the participant compile the data pertinent to the investigators primary and secondary outcomes. This diary should take no more than a minute or two for each sampling time. Participants will receive two phone calls at home to obtain this data at 8hrs and 24hrs.

ELIGIBILITY:
Inclusion Criteria:

* All patient's scheduled for elective unilateral open inguinal hernia repair at WFUBMC.

Exclusion Criteria:

* The anesthesiologist performing the intraoperative anesthetic deems the patient inappropriate for general anesthesia.
* If the patient uses more than 40mg of Oxycodone equivalents per 24 hours or is on extended release opioid formulations.
* If there is a contraindication to the performance of a regional block
* Concomitant anticoagulation use
* Allergy to local anesthetic
* Infectious or dermatologic conditions in the area of block placement that would otherwise increase the risk of peripheral nerve blockade
* Patient refusal
* Pregnancy
* Institutionalized individuals
* Extremes of age: Age > 90 or < 18
* Non English speaking

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2018-02-17 (Actual); Study Completion 2018-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Edwards, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Williams BA, Kentor ML, Vogt MT, Vogt WB, Coley KC, Williams JP, Roberts MS, Chelly JE, Harner CD, Fu FH. Economics of nerve block pain management after anterior cruciate ligament reconstruction: potential hospital cost savings via associated postanesthesia care unit bypass and same-day discharge. Anesthesiology. 2004 Mar;100(3):697-706. doi: 10.1097/00000542-200403000-00034. PMID 15108988
- [Background] Toivonen J, Permi J, Rosenberg PH. Analgesia and discharge following preincisional ilioinguinal and iliohypogastric nerve block combined with general or spinal anaesthesia for inguinal herniorrhaphy. Acta Anaesthesiol Scand. 2004 Apr;48(4):480-5. doi: 10.1111/j.1399-6576.2004.00346.x. PMID 15025612
- [Background] Børglum J, Jensen K, Moriggl B, et al. Ultrasound-Guided Transmuscular Quadratus Lumborum Blockade. BJA Out Blue E-Letters 2013. Available from http://bja.oxfordjournals. org/forum/topic/brjana_el%3B9919 (accessed 16 December 2015)
- [Background] Farrar JT, Berlin JA, Strom BL. Clinically important changes in acute pain outcome measures: a validation study. J Pain Symptom Manage. 2003 May;25(5):406-11. doi: 10.1016/s0885-3924(03)00162-3. PMID 12727037
- [Background] Willschke H, Marhofer P, Bosenberg A, Johnston S, Wanzel O, Cox SG, Sitzwohl C, Kapral S. Ultrasonography for ilioinguinal/iliohypogastric nerve blocks in children. Br J Anaesth. 2005 Aug;95(2):226-30. doi: 10.1093/bja/aei157. Epub 2005 May 27. PMID 15923270
- [Background] Schuirmann DJ. A comparison of the two one-sided tests procedure and the power approach for assessing the equivalence of average bioavailability. J Pharmacokinet Biopharm. 1987 Dec;15(6):657-80. doi: 10.1007/BF01068419. PMID 3450848
- [Background] 7. Julious SA. Sample Sizes for Clinical Trials. Chapman and Hall/CRC, Boca Raton, FL, 2010.

RESULTS

PARTICIPANT FLOW:
Groups:
- Quadratus Lumborum Block: Patient's randomized to receive a Quadratus Lumborum block (QLB) for post operative analgesia following inguinal herniorrhaphy will have said block performed in a lateral position in a manner consistent with the technique described by Børglum. Either a Sonosite linear HFL38x/13-6 MHz or Sonosite curvilinear C60x/5-2 MHz probe will be utilized to visualize the pertinent ultrasound anatomy. A Pajunk 21g x 100mm Sono Plex Stim Cannula will be utilized to appropriately deposit a single local anesthetic aliquot consisting of 25cc's of bupivacaine 0.25% with epinephrine 5mcg/cc and clonidine 1.66mcg/cc.
  Quadratus Lumborum Block: Patients randomized to this arm will receive 25cc's of Bupivacaine 0.25% + Epinephrine 1:200k + Clonidine 1.66mcg/cc administered via an ultrasound guided quadratus lumborum block technique.
  Bupivacaine 0.25%: Administered as part of the local anesthetic mixture Epinephrine 1:200k: Administered as part of the local anesthetic mixture Clonidine 1.66mcg/c
Period: Overall Study
Arm/Group | Ilioinguinal / Iliohypogastric Block | Quadratus Lumborum Block
Started | 30 | 30
Completed | 29 | 30
Not Completed | 1 | 0
Not completed — Did not meeting inclusion/exclusion | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ilioinguinal / Iliohypogastric Block | Quadratus Lumborum Block | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.4 (18.6) | 58.9 (11.2) | 56.2 (14.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 26 | 27 | 53
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 17 | 25 | 42
  African American | 10 | 4 | 14
  Hispanic | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 29 | 30 | 59
BMI [Median (Standard Deviation); unit: kg/m^2] | 25.2 (4.3) | 26.4 (6.2) | 25.8 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Verbal Pain Score With Movement
Description: Assessed on an 11-point (0-10) numeric analog scale with a higher score denoting a worse outcome.
Time Frame: 8 hrs Post Nerve Block
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ilioinguinal / Iliohypogastric Block | Quadratus Lumborum Block
Number analyzed (Participants) | 29 | 30
score on a scale | 5.10 (3.02) | 5.03 (3.01)

2. Secondary Outcome: Post-operative Verbal Pain Score at Rest
Description: Assessed on an 11-point (0-10) numeric analog scale with a higher score denoting a worse outcome
Time Frame: 8 hrs Post Nerve Block
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ilioinguinal / Iliohypogastric Block | Quadratus Lumborum Block
Number analyzed (Participants) | 29 | 30
score on a scale | 3.6 (3) | 3.3 (2.7)

3. Secondary Outcome: Post-operative Verbal Pain Score at Rest
Description: Assessed on an 11 point (0-10) numeric analog scale with a higher score denoting a worse outcome
Time Frame: 24 hrs Post Nerve Block
Population: One patient was lost to follow up in the Ilioinguinal Block arm after the 8 hour post block time point which is why the patient flow number for that arm differs from the 24 hour time frame.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ilioinguinal / Iliohypogastric Block | Quadratus Lumborum Block
Number analyzed (Participants) | 28 | 30
score on a scale | 3 (2.4) | 2.7 (2.2)

4. Secondary Outcome: Post-operative Verbal Pain Score With Activity
Description: Assessed on an 11 point (0-10) numeric analog scale with a higher score denoting a worse outcome
Time Frame: 24hrs Post Nerve Block
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ilioinguinal / Iliohypogastric Block | Quadratus Lumborum Block
Number analyzed (Participants) | 28 | 30
score on a scale | 4.9 (2.5) | 5.3 (2.4)

5. Secondary Outcome: Time to First Oral Analgesic
Description: When does the patient require their first post operative analgesic dose?
Time Frame: 24hrs Post Nerve Block
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Ilioinguinal / Iliohypogastric Block | Quadratus Lumborum Block
Number analyzed (Participants) | 28 | 30
minutes | 141 [71 to 742] | 91 [58 to 390]

6. Secondary Outcome: Time to Onset of Post Operative Pain
Description: When does the patient first note post operative pain?
Time Frame: 24hrs Post Nerve Block
Population: Data not collected
Arm/Group | Ilioinguinal / Iliohypogastric Block | Quadratus Lumborum Block
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Total Opioid Consumption
Description: Total opioids consumed during the first 24hrs post operatively. Measured as 24hr Oxycodone Equivalent
Time Frame: 24 hrs Post Nerve Block
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Ilioinguinal / Iliohypogastric Block | Quadratus Lumborum Block
Number analyzed (Participants) | 28 | 30
milligrams | 19.7 (19) | 25.2 (22)

8. Secondary Outcome: Number of Participants With Presence of Opioid Related Side Effects--Nausea
Time Frame: 8 hrs Post Nerve Block
Measure: Count of Participants; unit: Participants
Arm/Group | Ilioinguinal / Iliohypogastric Block | Quadratus Lumborum Block
Number analyzed (Participants) | 29 | 30
Participants | 9 | 5

9. Secondary Outcome: Number of Participants With Presence of Opioid Related Side Effects--Itching
Time Frame: 24 hrs Post Nerve Block
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Ilioinguinal / Iliohypogastric Block | Quadratus Lumborum Block
Number analyzed (Participants) | 28 | 30
Participants | 2 | 3

10. Secondary Outcome: Number of Participants With Presence of Opioid Related Side Effects--Itching
Time Frame: 8 hrs Post Nerve Block
Measure: Count of Participants; unit: Participants
Arm/Group | Ilioinguinal / Iliohypogastric Block | Quadratus Lumborum Block
Number analyzed (Participants) | 29 | 30
Participants | 0 | 4

11. Secondary Outcome: Number of Participants With Presence of Opioid Related Side Effects--Vomiting
Time Frame: 8 hrs Post Nerve Block
Measure: Count of Participants; unit: Participants
Arm/Group | Ilioinguinal / Iliohypogastric Block | Quadratus Lumborum Block
Number analyzed (Participants) | 29 | 30
Participants | 3 | 3

12. Secondary Outcome: Number of Participants With Presence of Opioid Related Side Effects--Nausea
Time Frame: 24 hrs Post Nerve Block
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Ilioinguinal / Iliohypogastric Block | Quadratus Lumborum Block
Number analyzed (Participants) | 28 | 30
Participants | 6 | 3

13. Secondary Outcome: Number of Participants With Presence of Opioid Related Side Effects--Vomiting
Time Frame: 24 hrs Post Nerve Block
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Ilioinguinal / Iliohypogastric Block | Quadratus Lumborum Block
Number analyzed (Participants) | 28 | 30
Participants | 3 | 2

ADVERSE EVENTS:
Time Frame: 8 - 24 hours
Arm/Group | Ilioinguinal / Iliohypogastric Block | Quadratus Lumborum Block
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 12/29 | 12/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ilioinguinal / Iliohypogastric Block (N=29) | Quadratus Lumborum Block (N=30)
Nausea (Gastrointestinal disorders) | 12 | 8
Vomiting (Gastrointestinal disorders) | 6 | 5
Itching (Skin and subcutaneous tissue disorders) | 2 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-18): https://cdn.clinicaltrials.gov/large-docs/66/NCT03007966/Prot_SAP_000.pdf